CLINICAL TRIAL: NCT00135902
Title: A Randomized Trial of Omega-3 Fatty Acid Supplementation to Prevent Preterm Birth in Pregnancies at High Risk
Brief Title: Omega-3 Fatty Acid Supplementation to Prevent Preterm Birth in High Risk Pregnancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HD36801-Omega-3; U10HD021410 (NIH); U10HD027869 (NIH); U10HD027917 (NIH); U10HD027860 (NIH); U10HD027915 (NIH); U10HD034208 (NIH); U10HD034136 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH); U10HD036801 (NIH)
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Progesterone; Omega-3 fatty acid; Pregnancy
MeSH Terms: conditions — Premature Birth | interventions — 17 alpha-Hydroxyprogesterone Caproate; 17-alpha-Hydroxyprogesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 17P plus Omega-3 Supplement (Active Comparator): Weekly 17 alpa hydroxyprogesterone caproate (17p) injections plus Omega 3 supplements, 4 capsules per day for up to 5 weeks. Each capsule contained 200 mg of docosahexaenoic acid (DHA) and 300 mg of eicosapentaenoic acid (EPA).
  Interventions: Drug: 17 alpha-Hydroxyprogesterone Caproate and Omega-3 supplement
- 17P plus Placebo Supplement (Placebo Comparator): Weekly 17 alpa hydroxyprogesterone caproate (17p) injections plus placebo capsules, 4 capsules per day for up to 5 weeks
  Interventions: Drug: 17 alpha-hydroxy progesterone caproate and Placebo supplement

INTERVENTIONS:
Drug: 17 alpha-Hydroxyprogesterone Caproate and Omega-3 supplement — Participants receive a weekly progesterone injection (17 alpha hydroxyprogesterone caproate) up to 37 weeks gestation and take daily Omega-3 supplements.
  Arms: 17P plus Omega-3 Supplement
Drug: 17 alpha-hydroxy progesterone caproate and Placebo supplement — Participants receive a weekly progesterone injection (17P) up to 37 weeks gestation and take daily placebo supplements
  Arms: 17P plus Placebo Supplement

SUMMARY:
A recently completed trial of weekly injections of 17 alpha hydroxyprogesterone caproate (17P) found significant effectiveness for 17P in preventing recurrent preterm birth. However, the group who received 17P in this trial still had a high rate of preterm birth. Several reports have shown that dietary supplementation of fish oil, which is rich in Omega-3 fatty acids, reduces the risk of preterm birth. This trial tests whether adding the Omega-3 supplement to 17P therapy has the potential for further reducing the risk of preterm birth in women who have previously had a spontaneous preterm delivery. The trial will compare Omega-3 fatty acid with placebo in women receiving 17P therapy. The hypothesis being tested is: "Among women at high risk for preterm birth receiving weekly injections of 17P, the addition of Omega-3 nutritional supplement will further reduce the rate of preterm birth."

DETAILED DESCRIPTION:
Preterm birth is the leading cause of perinatal mortality and morbidity. In a recently completed trial of weekly injections of 17 alpha hydroxyprogesterone caproate (17P), the National Institute of Child Health and Human Development (NICHD) Maternal Fetal Medicine Units (MFMU) Network found the treatments significantly beneficial in the prevention of recurrent preterm birth. Other studies have shown that fish oil supplementation can reduce the risk for preterm birth. The purpose of this study is to determine whether Omega-3, a polyunsaturated fatty acid nutritional supplement, in addition to injections of 17P, further decreases the rate of preterm birth in women at risk.

This study is a randomized, double-masked clinical trial with two study arms: a daily supplement of Omega-3 capsules containing 800 mg of DHA and 1200 mg of EPA or a daily supplement of a matching placebo. All patients will also receive weekly injections of 17P. Eight hundred pregnant women with a history of previous preterm delivery will be recruited for this study. After successfully completing a compliance run-in, which can begin as early as 15 weeks gestation, patients will be randomized and begin treatment between 16 and 22 weeks gestation. They will remain on study drug until 36 week and 6 days or delivery, whichever occurs first. Blood will be drawn at randomization and at a monthly visit falling between 25-29 weeks of gestation to test for compliance, to analyze genetic polymorphisms and to determine whether Omega-3 affects the production of inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of previous singleton spontaneous birth
* Singleton pregnancy
* Gestational age at randomization between 16 and 22 weeks

Exclusion Criteria:

* Major fetal anomaly or demise
* Regular intake of fish oil supplements
* Daily use of nonsteroidal anti-inflammatory agents
* Allergy to fish or fish products
* Gluten intolerant
* Heparin use or known thrombophilia
* Hemophilia
* Planned termination
* Current hypertension or current use of antihypertensive medications
* Type D, F or R diabetes
* Maternal medical complications
* Current or planned cerclage
* Illicit drug or alcohol abuse during current pregnancy
* Delivery at a non-Network hospital
* Participation in another pregnancy intervention study
* Participation in this trial in a previous pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2005-02; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Delivery before than 37 weeks gestation | Up to 37 weeks gestation
  Delivery before 37 weeks including any miscarriages occurring after randomization

SECONDARY OUTCOMES:
Delivery before 35 weeks gestation | Up to 35 weeks gestation
Delivery before 32 weeks gestation | Up to 32 weeks gestation
Delivery after 40 weeks gestation | 40 weeks gestation or greater
Pregnancy loss or neonatal death | Randomization to hospital discharge (up to 25 weeks)
Gestational age at delivery | Delivery
Birth weight less than 2,500 grams | Birth
Birth weight less than 1,500 grams | Birth
Birth size small for gestational age at less than 10th percentile | Birth
Birth size large for gestational age at more than 90th percentile | Birth
Admission to neonatal intensive care or intermediate care nursery | Delivery through neonatal discharge (up to 2 weeks)
Neonatal retinopathy of prematurity | Delivery through neonatal discharge (up to 2 weeks)
Intraventricular Hemorrhage at any grade | Delivery through neonatal discharge (up to 2 weeks)
Intraventricular Hemorrhage Grade 3 or 4 | Delivery through neonatal discharge (up to 2 weeks)
Neonatal patent ductus arteriosus | Delivery through neonatal discharge (up to 2 weeks)
Neonatal necrotizing enterocolitis | Delivery through neonatal discharge (up to 2 weeks)
Neonatal sepsis | Delivery through neonatal discharge (up to 2 weeks)
Neonatal respiratory distress syndrome | Delivery through neonatal discharge (up to 2 weeks)
Neonatal surfactant use | Delivery through neonatal discharge (up to 2 weeks)
Neonatal bronchopulmonary dysplasia | Delivery through neonatal discharge (up to 2 weeks)
Neonatal transient tacypnea | Delivery through neonatal discharge (up to 2 weeks)
Neonatal supplemental oxygen support | Delivery through neonatal discharge (up to 2 weeks)
Neonatal ventilator support | Delivery through neonatal discharge (up to 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Miodovnik, MD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Elizabeth A Thom, PhD, Principal Investigator — George Washington University Biostatistics Center; Margaret Harper, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (12):
- United States (12):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Wayne State University, Detroit, Michigan
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Case Western University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pittsburgh Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after completion and publication of the main analyses in accordance with NIH policy. The contact to obtain datasets is mfmudatasets@bsc.gwu.edu.

REFERENCES:
- [Background] Meis PJ, Klebanoff M, Thom E, Dombrowski MP, Sibai B, Moawad AH, Spong CY, Hauth JC, Miodovnik M, Varner MW, Leveno KJ, Caritis SN, Iams JD, Wapner RJ, Conway D, O'Sullivan MJ, Carpenter M, Mercer B, Ramin SM, Thorp JM, Peaceman AM, Gabbe S; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Prevention of recurrent preterm delivery by 17 alpha-hydroxyprogesterone caproate. N Engl J Med. 2003 Jun 12;348(24):2379-85. doi: 10.1056/NEJMoa035140. PMID 12802023
- [Background] Olsen SF, Secher NJ, Bjornsson S, Weber T, Atke A. The potential benefits of using fish oil in relation to preterm labor: the case for a randomized controlled trial? Acta Obstet Gynecol Scand. 2003 Nov;82(11):978-82. doi: 10.1034/j.1600-0412.2003.00334.x. No abstract available. PMID 14616269
- [Background] Duley L. Prophylactic fish oil in pregnancy. The Cochrane Pregnancy & Childbirth Database (Issue 2, 1995).
- [Background] Olsen SF, Secher NJ, Tabor A, Weber T, Walker JJ, Gluud C. Randomised clinical trials of fish oil supplementation in high risk pregnancies. Fish Oil Trials In Pregnancy (FOTIP) Team. BJOG. 2000 Mar;107(3):382-95. doi: 10.1111/j.1471-0528.2000.tb13235.x. PMID 10740336
- [Background] Olsen SF, Secher NJ. Low consumption of seafood in early pregnancy as a risk factor for preterm delivery: prospective cohort study. BMJ. 2002 Feb 23;324(7335):447. doi: 10.1136/bmj.324.7335.447. PMID 11859044
- [Background] Reece MS, McGregor JA, Allen KG, Harris MA. Maternal and perinatal long-chain fatty acids: possible roles in preterm birth. Am J Obstet Gynecol. 1997 Apr;176(4):907-14. doi: 10.1016/s0002-9378(97)70620-3. PMID 9125620
- [Background] Dunstan JA, Mori TA, Barden A, Beilin LJ, Taylor AL, Holt PG, Prescott SL. Fish oil supplementation in pregnancy modifies neonatal allergen-specific immune responses and clinical outcomes in infants at high risk of atopy: a randomized, controlled trial. J Allergy Clin Immunol. 2003 Dec;112(6):1178-84. doi: 10.1016/j.jaci.2003.09.009. PMID 14657879
- [Background] Cadroy Y, Dupouy D, Boneu B. Arachidonic acid enhances the tissue factor expression of mononuclear cells by the cyclo-oxygenase-1 pathway: beneficial effect of n-3 fatty acids. J Immunol. 1998 Jun 15;160(12):6145-50. PMID 9637532
- [Background] Lee JY, Plakidas A, Lee WH, Heikkinen A, Chanmugam P, Bray G, Hwang DH. Differential modulation of Toll-like receptors by fatty acids: preferential inhibition by n-3 polyunsaturated fatty acids. J Lipid Res. 2003 Mar;44(3):479-86. doi: 10.1194/jlr.M200361-JLR200. Epub 2002 Dec 1. PMID 12562875
- [Background] Calder PC. Dietary fatty acids and the immune system. Nutr Rev. 1998 Jan;56(1 Pt 2):S70-83. doi: 10.1111/j.1753-4887.1998.tb01648.x. No abstract available. PMID 9481127
- [Result] Harper M, Thom E, Klebanoff MA, Thorp J Jr, Sorokin Y, Varner MW, Wapner RJ, Caritis SN, Iams JD, Carpenter MW, Peaceman AM, Mercer BM, Sciscione A, Rouse DJ, Ramin SM, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Omega-3 fatty acid supplementation to prevent recurrent preterm birth: a randomized controlled trial. Obstet Gynecol. 2010 Feb;115(2 Pt 1):234-242. doi: 10.1097/AOG.0b013e3181cbd60e. PMID 20093894
- [Derived] Harper M, Li L, Zhao Y, Klebanoff MA, Thorp JM Jr, Sorokin Y, Varner MW, Wapner RJ, Caritis SN, Iams JD, Carpenter MW, Peaceman AM, Mercer BM, Sciscione A, Rouse DJ, Ramin SM, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Change in mononuclear leukocyte responsiveness in midpregnancy and subsequent preterm birth. Obstet Gynecol. 2013 Apr;121(4):805-811. doi: 10.1097/AOG.0b013e3182878a80. PMID 23635681
- [Derived] Klebanoff MA, Harper M, Lai Y, Thorp J Jr, Sorokin Y, Varner MW, Wapner RJ, Caritis SN, Iams JD, Carpenter MW, Peaceman AM, Mercer BM, Sciscione A, Rouse DJ, Ramin SM, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). Fish consumption, erythrocyte fatty acids, and preterm birth. Obstet Gynecol. 2011 May;117(5):1071-1077. doi: 10.1097/AOG.0b013e31821645dc. PMID 21508745
- [Derived] Harper M, Zheng SL, Thom E, Klebanoff MA, Thorp J Jr, Sorokin Y, Varner MW, Iams JD, Dinsmoor M, Mercer BM, Rouse DJ, Ramin SM, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). Cytokine gene polymorphisms and length of gestation. Obstet Gynecol. 2011 Jan;117(1):125-130. doi: 10.1097/AOG.0b013e318202b2ef. PMID 21173653
- See also: Related Info — http://www.bsc.gwu.edu/mfmu